CLINICAL TRIAL: NCT02231957
Title: Text Message Vaccine Reminders for Adolescents With Chronic Medical Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Annika Hofstetter, Assistant Professor of Pediatrics, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: AAAM3756
Record Dates: First submitted 2014-08-15; First posted 2014-09-04 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Vaccination

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- educational text message reminders (Experimental): receipt of education-embedded text message vaccine reminders
  Interventions: Other: educational text message reminders
- conventional text message reminders (Active Comparator): receipt of conventional text message vaccine reminders
  Interventions: Other: conventional text message reminders

INTERVENTIONS:
Other: educational text message reminders
  Other Names: educational text message vaccine reminders; education-embedded text message vaccine reminders
  Arms: educational text message reminders
Other: conventional text message reminders
  Other Names: conventional text message vaccine reminders
  Arms: conventional text message reminders

SUMMARY:
There are a growing number of adolescents with chronic medical conditions in the United States. The Advisory Committee on Immunization Practices (ACIP) recommends HPV vaccination and annual influenza vaccination of all adolescents. Pneumococcal polysaccharide vaccination is also recommended for certain high-risk patients. Limited studies suggest that vaccination coverage of this population remains sub-optimal. Text message vaccine reminder/recall has been shown to be effective in increasing uptake of select pediatric and adolescents vaccines, but has yet to be examined among patients with chronic medical conditions who may also face unique barriers to vaccination. This intervention aims to implement and evaluate the use of text message vaccine reminders among urban low-income minority adolescents with chronic medical conditions. This investigator-initiated study is supported in part by a grant from the Pfizer Medical Education Group.

ELIGIBILITY:
Inclusion Criteria:

Parent with

1. adolescent aged 11-17 years;
2. adolescent with ≥1 chronic medical condition;
3. adolescent with clinic visit in last 12 months;
4. cell phone number listed in hospital registration system

Exclusion Criteria:

Parent who:

1. does not speak English or Spanish;
2. is unwilling to receive text message vaccine reminders;
3. anticipates moving from area in coming 12 months

Min Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Percentage of eligible subjects who received HPV1, influenza, and/or pneumococcal vaccine(s) | 12 weeks after intervention start

SECONDARY OUTCOMES:
Percentage of eligible subjects who received HPV1, influenza, and/or pneumococcal vaccine(s) | 4 weeks after intervention start
Percentage of eligible subjects who received HPV1, influenza, and/or pneumococcal vaccine(s) | 24 weeks after intervention start
Percentage of eligible subjects with missed opportunities for HPV1, influenza, and/or pneumococcal vaccination | 4 weeks after intervention start
Percentage of eligible subjects with missed opportunities for HPV1, influenza, and/or pneumococcal vaccination | 12 weeks after intervention start
Percentage of eligible subjects with missed opportunities for HPV1, influenza, and/or pneumococcal vaccination | 24 weeks after intervention start

CONTACTS AND LOCATIONS:
Overall Officials: Annika M Hofstetter, MD, PhD, MPH, Principal Investigator — Columbia University
Locations (1):
- NewYork-Presbyterian Hospital/Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Derived] Hofstetter AM, Barrett A, Camargo S, Rosenthal SL, Stockwell MS. Text message reminders for vaccination of adolescents with chronic medical conditions: A randomized clinical trial. Vaccine. 2017 Aug 16;35(35 Pt B):4554-4560. doi: 10.1016/j.vaccine.2017.07.022. Epub 2017 Jul 21. PMID 28736201